CLINICAL TRIAL: NCT05345717
Title: Novel Desensitization Protocol With Proteasome Inhibitor and Costimulation Blockade for Highly Sensitized Patients to Allow for Successful Kidney Transplantation. A Pilot Study.
Brief Title: Novel Desensitization Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0323
Record Dates: First submitted 2021-12-03; First posted 2022-04-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplantation; End Stage Kidney Disease (ESRD)
Keywords: kidney transplantation; sensitized patients; belatacept; proteasome inhibitor
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Abatacept; Proteasome Inhibitors

STUDY DESIGN:
Intervention Model Description: A pilot study on 5 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients treated with belatacept and proteasome inhibitor (Experimental): Highly sensitized patients will be treated with belatacept and proteasome inhibitor and monitored for decreasing calculated Panel of Reactive Antibodies (cPRA) and suitable kidney donor base don negative crossmatch
  Interventions: Drug: Belatacept Injection

INTERVENTIONS:
Drug: Belatacept Injection — Patient will initiate belatacept therapy and will received 2 cycles of proteasome inhibitor therapy
  Other Names: proteasome inhibitor

SUMMARY:
This proposal's objective is to determine whether belatacept, in conjunction with a proteasome inhibitor can be used to safely increase the likelihood of finding an acceptable donor for highly HLA sensitized kidney transplant candidates.

DETAILED DESCRIPTION:
This is a pilot study to test the safety and effectiveness of the desensitization therapy with belatacept and proteasome inhibitor to increase the likelihood of of finding an acceptable donor for highly HLA sensitized kidney transplant candidates.

ELIGIBILITY:
Inclusion Criteria:

* Highly sensitized patient cPRA 99-100% AND actively listed for kidney transplantation at the kidney transplantation Program at University fo Chicago
* Ebstein Barr Virus (EBV) Immunoglobulins (IgG) seropositive
* No active systemic infection
* No allergy to proteasome inhibitors (Bortezomib), or to belatacept
* No known malignancy in the previous 2 years except for non-melanomatous skin cancer
* Female who agrees to practice 2 effective methods of contraception through 3 months after the last dose of Bortezomib
* Patient vaccinated against hepatitis B virus with positive level of HBsAb
* Patients fully vaccinated against Coronavirus Disease 2019 at least 2 weeks prior to the start of the 1st cycle.
* Actively listed for kidney transplant at the Transplant Institute at University of Chicago

Exclusion Criteria:

* Patient with significant neuropathy by the Common Terminology Criteria for Adverse Events (CTCAE) criteria within 14 days before enrollment (Grades 3-4 or Grade 2 with pain)
* Myocardial infarction within 6 months of enrollment or has Heart Failure in acute dialysis quality initiative (ADQI) ESRD classification system Class 2 non restrictive (2NR) or greater, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities
* Patient who received other investigational drugs within 14 days prior to initiation of study treatment
* Receipt of a live vaccine within 4 weeks prior to initiation of study treatment
* Evidence of severe liver disease by history or physical exam or with abnormal liver profile ( > 1.5 times upper limit of normal within 30 days of consent)
* Female who is breast feeding or pregnant
* Untreated latent tuberculosis
* History of Post Transplant Lymphoproliferative Disease (PTLD)
* Patient still carrying previous kidney transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Likelihood of finding a donor to whom the study participant does not have strong anti-donor HLA specific antibodies (DSA). | 1 year
  The likelihood of finding a suitable donor will calculated base on calculated Panel of Reactive Antibodies measured 1month after the therapy

SECONDARY OUTCOMES:
Strong Human Leukocyte Antigen (HLA) antibodies with mean fluorescence intensity (MFI) reduced by more than 50% | 1 year
  A number of strong HLA antibodies with MFI reduced by more than 50% will be counted
Time to transplant | 1 year
  Time from the beginning of the implementation of the therapy to kidney transplantation will be measured
Episodes of Antibody Mediated Rejection (AMR) and Acute Cellular Rejection (ACR) | 1 year
  Number of episodes of AMR and ACR after kidney transplantation will be counted
Death | 1 year
  The incidence of episodes of patient death will be calculated
Serious infection requiring inpatient intravenous therapies | 1 year
  Incidence rate of the episodes of serious infection requiring inpatient intravenous therapies will be calculated during the study
Post-transplant lymphoproliferative disorder | 1 year
  The incidence rate of the episodes of post-transplant lymphoproliferative disorder will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Witkowski, MD PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States